CLINICAL TRIAL: NCT07261137
Title: A Randomized, Controlled Clinical Study Evaluating the Efficacy of Solventum™ Vitrebond™ Pulp Protect Liner/Base Used as a Liner/Base Under Dental Restorations
Brief Title: Efficacy of Solventum™ Vitrebond™ Pulp Protect Liner/Base Used as a Liner/Base Under Dental Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EM-11-050090
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Caries, Dental; Tooth Decay; Dental Decay; Tooth Sensitivity
Keywords: dental; caries; liner-base; tooth sensitivity; Vitrebond Pulp Protect; Vitrebond Plus; pulp vitality
MeSH Terms: conditions — Dental Caries; Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: randomized, controlled, partially blinded, clinical study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vitrebond™ Pulp Protect Liner/Base (Experimental): Study tooth will be treated with Vitrebond™ Pulp Protect Liner/Base as a liner/base.
  Interventions: Device: Vitrebond™ Pulp Protect Liner/Base
- Vitrebond™ Plus (Active Comparator): Study tooth will be treated with Vitrebond™ Plus (comparator) as a liner/base.
  Interventions: Device: Vitrebond™ Plus (comparator)

INTERVENTIONS:
Device: Vitrebond™ Pulp Protect Liner/Base — Vitrebond™ Pulp Protect Liner/Base used as a liner / base during restoration of permanent teeth with moderate or advanced occlusal and/or proximal caries.
  Arms: Vitrebond™ Pulp Protect Liner/Base
Device: Vitrebond™ Plus (comparator) — Vitrebond™ Plus used as a liner / base during restoration of permanent teeth with moderate or advanced occlusal and/or proximal caries.
  Arms: Vitrebond™ Plus

SUMMARY:
This is a clinical study evaluating a new dental product called Solventum™ Vitrebond™ Pulp Protect Liner/Base. This new product is designed to be used as a liner or base between the tooth and the dental filling, as well as for a procedure called direct pulp capping (DPC) if there is exposed pulp. Dental pulp is the part of the tooth that contains the nerves, blood vessels, and cells that keep your tooth healthy. This study will focus specifically on the liner/base application.

In this study, the Solventum study product will be compared to a similar, commercially available product made by Solventum called 3M™ Vitrebond™ Plus Light Cure Glass Ionomer Liner/Base (Vitrebond Plus for short). The study will include participants who are at least 7 years old who have at least one tooth with moderate or advanced caries (tooth decay).

The entire duration of the study is anticipated to be 2 years from when the first subject begins the study until the last subject completes the study. The duration of each study subject's participation will be up to 1 year consisting of an initial tooth restoration visit at baseline, a subject self-reported post-operative sensitivity assessment at 1 week reported by phone call, and in-person follow-up assessments at 1 month, 6 months, and 1 year post-restoration to confirm safety and effectiveness. The study will be partially blinded, which means that the participant and the dentist doing the assessments won't know which liner/base product is used on their tooth.

DETAILED DESCRIPTION:
This is a single-site, randomized, controlled, partially blinded, non-inferiority, parallel-group study comparing two liner/base materials: Solventum™ Vitrebond™ Pulp Protect Liner/Base and 3M™ Vitrebond™ Plus. Both products will be used as intended in accordance with their cleared labeling. Restorations on study teeth will be performed in accordance with the relevant manufacturer's Instructions for Use and the clinical investigation plan.

Enough Subjects will be enrolled and confirmed eligible to treat 128 teeth with either Vitrebond Pulp Protect or Vitrebond Plus (64 per treatment arm) as the liner/base. A single eligible tooth with moderate or advanced occlusal and/or proximal caries per subject may be included in the study. Randomization will be stratified by caries depth as determined during screening such that there will be a targeted 1:1 ratio of the two treatment arms allocated for each stratum. There will be no minimum size requirement for enrollment by caries depth.

Intra-oral photographs will be taken of the prepared tooth on the day of restoration just prior to and just after lining/basing the cavity floor. Standard dental radiographs (x-rays) will be taken at baseline for the screening purposes to determine tooth eligibility.

Tooth sensitivity assessments will be self-reported by subjects. All other assessments will be performed by dental examiners who are independent of the dentist who performed the restoration procedure and are blinded to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 7 years of age or older at time of consent.
2. Subject or Subject's Legally Authorized Representative is able to understand and willing to sign an Informed Consent Form or give Assent, as applicable.
3. Subject is able and willing to attend all scheduled study visits.
4. Subject is able and willing to follow study restrictions.
5. Subject is in good general health (i.e., meets ASA Level I or ASA Level II classification criteria).
6. Subject has at least 1 permanent tooth with moderate or advanced (per ICDAS Guidelines/ADA caries classification system) occlusal and/or proximal caries based upon clinical and/or radiographic evaluation.
7. Subject has existing dental radiographic images of acceptable diagnostic quality taken within 1 month of tooth restoration.
8. Study tooth has healthy periodontal tissues or mildly inflamed tissues, with probing depths no greater than 4 mm and no gingival recession associated with self-reported sensitivity.
9. Study tooth has a positive response to a sensibility test (i.e., cold test using a refrigerant spray).
10. Study tooth has no pre-operative sensitivity or exhibit pre-operative sensitivity that is relieved immediately after stimulus removal.
11. Study tooth can be restored with a direct permanent restoration (stepwise caries removal will not be used).
12. Study tooth involving multiple carious surfaces can be restored with a single, continuous restoration (excluding buccal and lingual surfaces).

Exclusion Criteria:

1. Subject has a history of adverse reaction to any materials used in this study, including but not limited to acrylates.
2. Subject is unable, for any reason, to tolerate the study procedures or the length of time required to complete the restoration(s) on the study tooth.
3. Subject is taking part in or planning to be enrolled in a clinical evaluation of any other dental materials at any time during the study.
4. Subject has a history of chronic use of anti-inflammatory, analgesic (pain), and/or mind-altering drugs for medical (including psychiatric) and pharmacotherapeutic therapies that might alter perception of pain.
5. Subject is pregnant or breast feeding at the time of screening.
6. Subject has any spontaneous or other orofacial pain (including toothache, percussion tenderness, and periapical radiolucency).
7. Subject has caries or conditions involving non-study teeth that may interfere with the sensitivity assessments (e.g., advanced caries in a non-study tooth in the same quadrant as the study tooth).
8. Subject has Temporal Mandibular Disorder with pain.
9. Study tooth with current or previous trauma or previous restorations.
10. Study tooth diagnosed with cracked tooth syndrome.
11. Study tooth with mobility >= grade 2 using the Miller's tooth mobility index.
12. Study tooth has previous and/or current signs or symptoms of pulpal and/or periapical disease (e.g., root resorption or pulpal calcifications) or irreversible pulpitis.
13. Tooth surface loss (attrition, erosion, abrasion or abfraction) on study tooth or adjacent teeth that could impact perception of pain.
14. Study tooth has no systemic mineralization pathology (e.g., amelogenesis imperfecta, enamel hypoplasia, etc).
15. Subject is, in the opinion of the Investigator, unsuitable for enrollment in the study for reasons other than those specified in the above exclusion criteria.

    Intra-Operative Exclusion Criteria:
16. Study tooth with pulp exposure under any circumstance (caries exposure, mechanical/traumatic).

Ages: 7 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Patient self-reported post-operative sensitivity at 1 week | 1 week
  Tooth sensitivity will be self-reported by subjects prior to tooth restoration to establish baseline, and post-operatively at 1 week post-restoration. Categories for pre/post-operative sensitivity will be graded on the following scale:
  1. Absence of pain/sensitivity
  2. Mild to moderate pain/sensitivity
  3. Severe / Spontaneous pain
  Spontaneous pain is defined as prolonged intense pain that doesn't respond to pain medication, and/or pain that wakes you up from sleep.

SECONDARY OUTCOMES:
Pulp Vitality | assessed at baseline, 1 month, 6 months, and 1 year after tooth restoration
  Pulp vitality assessed by pulp sensibility testing response to cold stimuli (i.e., endo ice). Pulp sensibility testing will be administered at baseline (pre-restoration), 1 month, 6 months, and 1 year post-procedure using a refrigerant spray intended for dental use. A positive response from the pulp sensibility test at the timepoints described is indicative of the pulp vitality of the tooth. A lower score is desired.
  Categories for pulp vitality will include:
  1. Vital pulp (normal): Positive response from the pulp sensibility test that subsides within 5 seconds.
  2. Reversible pulpitis: Positive response from pulp sensibility test that lasts greater than 5 seconds up to 30 seconds.
  3. Irreversible pulpitis: Prolonged positive response from pulp sensibility test that lasts more than 30 seconds.
  4. Non-vital pulp: Negative response from the pulp sensibility test.
Patient self-reported post-operative sensitivity at 1 month | 1 month
  Tooth sensitivity will be self-reported by subjects prior to tooth restoration to establish baseline, and post-operatively at 1 month post-restoration. Categories for pre/post-operative sensitivity will be graded on the following scale:
  1. Absence of pain/sensitivity
  2. Mild to moderate pain/sensitivity
  3. Severe / Spontaneous pain
  Spontaneous pain is defined as prolonged intense pain that doesn't respond to pain medication, and/or pain that wakes you up from sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Mabi Singh, DMD, BDS, MS, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No